CLINICAL TRIAL: NCT04325724
Title: Monocentric Cross-sectional Study Assessing the Role of Inflammatory and Structural Ultrasound Abnormalities by Explaining the Perspective of Patients With Psoriatic Arthritis
Brief Title: Evaluation of the Role of Inflammatory and Structural Ultrasound Abnormalities by Explaining the Perspective of Patients With Psoriatic Arthritis
Acronym: EchoPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP 190620; 2019-A01839-48 (Other: IDRCB)
Record Dates: First submitted 2020-02-17; First posted 2020-03-30 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-02

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Who Masked: Investigator
Masking Description: ultrasound evaluation will be on masking from clinical evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Beginner psoriatic arthritis patients (Other): Every patients consulting in dermatologic or rheumatologic department for a skin psoriasis with clinical symptoms which may lead to the suspicion of psoriatic arthritis
  Interventions: Other: General evaluation; Other: Dermatological evaluation; Other: Rheumatological evaluation; Other: para clinical data; Other: Patient reported outcomes (PROs)
- Confirmed psoriatic arthritis patients (Other): Every patients with psoriatic arthritis followed in rheumatologic department
  Interventions: Other: General evaluation; Other: Dermatological evaluation; Other: Rheumatological evaluation; Other: para clinical data; Other: Patient reported outcomes (PROs)
- Rheumatoid arthritis or Digital osteoarthritis patients (Other): Followed in rheumatologic department
  Interventions: Other: General evaluation; Other: Rheumatological evaluation; Other: para clinical data; Other: Patient reported outcomes (PROs)
- Skin psoriasis patients without any articular symptoms (Other)
  Interventions: Other: General evaluation; Other: Dermatological evaluation; Other: Rheumatological evaluation; Other: para clinical data; Other: Patient reported outcomes (PROs)

INTERVENTIONS:
Other: General evaluation — Demographic characteristic, psoriasis duration, disease duration, treatments
Other: Dermatological evaluation — treatment and evaluation
  Arms: Beginner psoriatic arthritis patients; Confirmed psoriatic arthritis patients; Skin psoriasis patients without any articular symptoms
Other: Rheumatological evaluation — joints, enthesis, tendons, and other ultrasound abnormalities
Other: para clinical data — biological data, medical imaging data
Other: Patient reported outcomes (PROs) — Psoriatic arthritis impact of disease 12 (PsAID12), hospital anxiety and depression scale (HAD), SF 36

SUMMARY:
The perspective of the patient is defined by the patient reported outcomes (PROs). This is a main part of the care in psoriatic arthritis. However , PROs can be influenced by environmental parameters.

Ultrasound represents an objective instrument in the context of psoriatic rheumatism (RhPso) care because it measures inflammatory activity and structural damage at joint and periarticular level.

it is the first study to evaluate the role of inflammatory and structural ultrasound abnormalities as a cause of modification of the patient's perspective measured by PROs in patients with RhPso.

DETAILED DESCRIPTION:
It is an interventional study. Patients will be enrolled in the rheumatology department Of Ambroise Paré Hospital in collaboration with the dermatology departments of the hospital.

All patients with psoriatic arthritis, beginner or established, or patients with psoriasis suspecting the beginning of rheumatism who will consult or are already followed in those departments and give their approval for the study will undergo

* a clinical rheumatologic assessment (number of painful or swollen joints, enthesitic pain, inflammatory spinal pain)
* an ultrasound assessment (peripheral joints, tendon and enthesitic structures and nails).

Those assessment will be made the same day of their consult in one those departments. They will be asked to complete questionnaires (PROs) on the overall assessment of the disease, pain, quality of life, tiredness, physical limitation / disability and the impact of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders above 18 years old
* Capable of adhering to the protocol
* Consent given
* Present one of those disease:
* RhPso (confirmed diagnosis) according to The Classification for Psoriatic arthritis criteria (CASPAR)
* Rheumatoid arthritis according to ACR/EULAR criteria (American College of Rheumatology/ European League Against Rheumatism)
* Digital osteoarthritis according to american college of rheumatology (ACR) criteria
* Cutaneous psoriasis
* Having signed a consent form
* Affiliated to a regimen of health insurance

Exclusion Criteria:

* Patient refusing the study
* The association of two rheumatic diseases (for example: psoriatic arthritis and gout, rheumatoid arthritis and arthritis etc)
* The association of another chronic pathology likely to lead to joint manifestations (systemic diseases, bowel chronic inflammatory diseases, overload diseases, ...)
* Patient under trusteeship or protection of vulnerable adults
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of patient global assessment (PGA) in patients with Psoriatic Arthritis | 1 day
  The study of patient global assessment will permit to understand the impact of inflammation and external structural damage measured by ultrasound in patients with psoriatic arthritis (newly diagnosed or with confirmed diagnosis).
  At enrollment visit (only visit) of patient PGA will be assessed with a digital scale from 0 to 10

SECONDARY OUTCOMES:
Evaluation of the impact of inflammation and external structural damage measured by ultrasound | 1 day
  Evaluate the impact of inflammation and external structural damage measured by ultrasound to explain the others PROs: PGA joint damage activity and cutaneous damage will be measure with a digital scale
Evaluation of the impact of inflammation and external structural damage measured by ultrasound | 1 day
  Evaluate the impact of inflammation and external structural damage measured by ultrasound to explain the others PROs: Pain will be assessed with a digital scale
Evaluation of the impact of inflammation and external structural damage measured by ultrasound | 1 day
  Evaluate the impact of inflammation and external structural damage measured by ultrasound to explain the others PROs: Physical limitation/ disability will be assessed with the health assessment questionnaire (HAQ)
Evaluation of the impact of inflammation and external structural damage measured by ultrasound | 1 day
  Evaluate the impact of inflammation and external structural damage measured by ultrasound to explain the others PROs: Quality of life will be assessed with a short form-36 (SF-36) questionnaire
Evaluation of the impact of inflammation and external structural damage measured by ultrasound | 1 day
  Evaluate the impact of inflammation and external structural damage measured by ultrasound to explain the others PROs: Disease effect will be assessed with psoriatic arthritis impact of disease (PsAID) 12 questionnaire
Evaluation of the impact of inflammation and external structural damage measured by ultrasound | 1 day
  Evaluate the impact of inflammation and external structural damage measured by ultrasound to explain the others PROs: Fatigue will be assessed with a digital scale
Evaluation of the impact of inflammation and external structural damage measured by ultrasound | 1 day
  Compare the results( prevalence of ultrasound irregularity, PROs, and factor which explain PROs) to people who suffer from psoriatic, without damage, without sign of joints damages or rheumatoid arthritis (RA) or digital osteoarthritis.
  Ultrasound damages: Synovitis, tenosynovitis, enthesitis, dactylitis, erosions, periosteal appositions ( enthesophytes, osteophyte and bony cortical irregularity) will be defined according to established by outcome measures in rheumatology (OMERACT) definitions and rating according to scores established by OMERACT

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Antonietta D'AGOSTINO, PhD, Principal Investigator — Rheumatology Department, Ambroise Paré Hospital

IPD SHARING:
Plan to Share IPD: No